CLINICAL TRIAL: NCT07110285
Title: Ovarian Stimulation Outcomes During a GnRH Antagonist Protocol for In-vitro Fertilization When Comparing Trigger Day Decision by Physicians Versus an Artificial Intelligence-based Algorithm - A Randomized Control Study.
Brief Title: Ovarian Stimulation Outcomes During a GnRH Antagonist Protocol for In-vitro Fertilization When Comparing Trigger Day Decision by Physicians Versus an Artificial Intelligence-based Algorithm.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FertilAI (Industry)
Responsible Party: Principal Investigator, Michal Youngster, Principal Investigator, FertilAI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0015-23-HMC
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-05

CONDITIONS: IVF Outcomes
Keywords: Trigger day decision; In-vitro fertilization; Mature oocytes; Artifical intelligence-based algorithm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician-based trigger day timing decision (No Intervention): Trigger day timing is decided on by the treating physician
- Artificial intelligence-based algorithm trigger day timing decision (Experimental): Trigger day timing decision by an artificial intelligence-based algorithm
  Interventions: Other: Artificial intelligence-based algorithm

INTERVENTIONS:
Other: Artificial intelligence-based algorithm — Trigger day timing decision by an artificial intelligence-based algorithm
  Arms: Artificial intelligence-based algorithm trigger day timing decision

SUMMARY:
To compare the number of mature oocytes following a GnRH antagonist in-vitro fertilization stimulation cycle when comparing trigger day timing decision by physicians versus an artificial intelligence-based algorithm

DETAILED DESCRIPTION:
Examination of all patients undergoing an ovarian stimulation cycle utilizing the GnRH antagonist protocol for oocyte cryopreservation or for fertilization via intracytoplasmic sperm injection (ICSI) (any treatment where oocytes are denuded and maturity may be assessed). The number of mature oocytes will be compared between cycles where trigger day timing was decided by the treating physician versus an artificial intelligence-based algorithm.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an ovarian stimulation cycle utilizing the GnRH antagonist protocol for oocyte cryopreservation or for fertilization via intracytoplasmic sperm injection (ICSI) (any treatment where oocytes are denuded and maturity may be assessed).

Exclusion Criteria:

* Loss to follow-up, patient retracts consent to participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Mature oocyte yield | 2 years
  The number of mature oocytes collected during a single egg retrieval cycle

SECONDARY OUTCOMES:
Oocyte yield | 2 years
  Number of retrieved oocytes during an egg collection cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Hourvitz, MD, Principal Investigator — Herzeliya Medical Center, Israel
Locations (1):
- Herzliya Medical Center, Herzliya, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data regarding patient demographics, characteristics and cycle outcomes (anynomized)
Supporting Information: Study Protocol
Time Frame: From the beginning until the end of recruitment